CLINICAL TRIAL: NCT00111254
Title: The Effects of Microdermabrasion on Collagen and Elastin Biosynthesis
Brief Title: The Effects of Microdermabrasion on Skin Remodeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Darius J. Karimipour, M.D., Clinical Assistant Professor, University of Michigan Department of Dermatology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Derm 486
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Skin; Skin Wrinkling
Keywords: microdermabrasion; skin; wrinkles; collagen; photoaging; wrinkled skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): In group I, acute effect group, each subject will undergo microdermabrasion of the hip/buttock. Treatment will consist of 3 passes in different directions (horizontal, vertical and oblique) with the microdermabrasion handpiece (Parisian Peel, Prestige model, medical microdermabrasion device). 4mm punch biopsies will be performed in the treated area at 4hrs, 8hrs, and 24hrs post-treatment. In addition, one 4mm punch biopsy will be obtained from adjacent untreated skin.
  Interventions: Procedure: Microdermabrasion
- 2 (Experimental): In group II, chronic effect group, each subject will undergo microdermabrasion of the face at weekly intervals for six weeks. Treatment will consist of 3 passes in different directions with the microdermabrasion handpiece (horizontal, vertical, and oblique). Aluminum oxide abrasion and negative pressure will be increased as tolerated by the patient. Two 2mm punch biopsies will be obtained prior to the first treatment and one week following the sixth treatment.
  Interventions: Procedure: Microdermabrasion

INTERVENTIONS:
Procedure: Microdermabrasion — Treatment will consist of 3 passes in different directions (horizontal, vertical and oblique) with the microdermabrasion handpiece (Parisian Peel, Prestige model, medical microdermabrasion device).

SUMMARY:
This research project aims to study the effects of microdermabrasion, a technique causing minimal injury used to improve the appearance of fine lines, wrinkles, and scars. Subjects will undergo microdermabrasion, which is a gentle "sand-blasting" of the skin. We are interested in determining how this procedure works at rebuilding the skin following microdermabrasion.

DETAILED DESCRIPTION:
Microdermabrasion is rapidly becoming one of the most popular cosmetic procedures performed by dermatologists and plastic surgeons. Microdermabrasion is a process that uses a high-pressure stream of aluminum oxide crystals and negative pressure to superficially peel the upper layer of the skin. Its purported benefits include improvement of photoaged skin, acne, and facial scarring.

The appeal of microdermabrasion is its effectiveness, simplicity, low patient and operator risk, and rapid recovery. Clinically, studies have illustrated beneficial effects on photodamaged skin.

Histologically, microdermabrasion has reproducible effects on the epidermis and dermis. Studies have shown a consistent increase in epidermal thickness as well as changes in the elastin content of the dermis while changes in collagen content have not been observed.

The reported clinical and histologic changes seen in previous studies suggest that alterations in the dermis precipitated by epidermal injury may be responsible for the beneficial effects of microdermabrasion on photoaging and scarring. In fact, others have reported that skin fibroblasts under tension may increase collagen synthesis.

Disruption of the epidermal barrier initiates a repair process that restores barrier function within hours to days, depending on the severity of the damage. This repair process involves increased synthesis of barrier lipids, followed by formation of new corneocytes. Elevated lipid synthesis largely occurs as a result of increased gene expression of the major enzymes responsible for lipid biosynthesis.

In this study, subjects will be assigned to one of two treatment groups. Patients in the first group will have their hip/buttock or forearm treated with the microdermabrasion machine. There may be only one treatment or as many as 6 on the same area, spaced up to two weeks apart. The treated area will be on either the right or left buttock and/or forearm and/or underarm. An area of approximately 10x10 cm (4x4 inches) will be treated. Skin biopsies will be performed on up to nine different times, up to six months following dermabrasion, on treated and/or untreated skin from the buttocks, forearm and/or underarm. Therefore, a total of (up to) nine biopsies will be taken from subjects in this group. The biopsies will be 4 mm or smaller in size, or about the size of a pencil eraser. Subjects can expect to make six visits to the hospital over a 3-4 week period of time.

Subjects assigned to the second group will have their face treated with microdermabrasion at a weekly to biweekly interval for a total of six treatments. One pair of biopsies will be taken prior to the first treatment, and the 2nd and 3rd pair will be taken on two different occasions no later than 3 months following the final treatment. Thus, the maximum number of biopsies in group II is six. The biopsies will be 2mm punch, "cookie-cutter", biopsies and will be taken from in front of the ear. Subjects can expect to make 8-10 visits to the hospital over a 2-3 month period of time.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Patients must be available for follow up visits for biopsies to comply with the requirements of the protocol.
* Patients must sign and understand the informed consent prior to participation in the study.
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study

Exclusion Criteria:

* Oral retinoid (vitamin-A like drugs) use within one year of entry into the study
* Topical retinoid use within 3 months of the study
* Patients with a history of excessive scarring
* Patients with significant medical history or concurrent illness which investigators feel is not safe for study participation
* Patients who have had any type of facial rejuvenation procedure or treatment (such as Botox injections, collagen implants, or chemical peels) within the past six months
* Non-compliant patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2002-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Observing changes over time with respect to the following biochemical endpoints: Procollagen I and III, matrix metalloproteinases (MMPs 1, 3, and 9), and several cytokines including Interleukins and Tumor Necrosis Factor. | Group I: 1-4 weeks; Group II: 1-3 months

SECONDARY OUTCOMES:
Changes in clinical features associated with sun-damaged or wrinkled skin. | Group I: 1-4 weeks, Group II: 1-3 months

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan

REFERENCES:
- [Derived] Karimipour DJ, Rittie L, Hammerberg C, Min VK, Voorhees JJ, Orringer JS, Sachs DL, Hamilton T, Fisher GJ. Molecular analysis of aggressive microdermabrasion in photoaged skin. Arch Dermatol. 2009 Oct;145(10):1114-22. doi: 10.1001/archdermatol.2009.231. PMID 19841398